CLINICAL TRIAL: NCT00730457
Title: A Two Part Study to Investigate the Safety and Immunogenicity of the VAX125 Influenza Vaccine in Healthy Adults Age 18-49 Years Part I: Phase I, Open-Label, Escalating Dose-Ranging Study Part II: Phase II, Double-Blind Placebo-Controlled Study
Brief Title: Phase 1 Safety and Immunogenicity Study in Healthy Adults of VAX125, a Recombinant HA-flagellin Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAX125-01
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: influenza; recombinant; hemagglutinin; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Intramuscular (i.m.) vaccination of a single dose of 0.1 µg, 0.3 µg, 1 µg, 2 µg, 3 µg, 5 µg and 8 µg of STF2.HA1 (SI) (VAX125).
  Interventions: Biological: VAX125

INTERVENTIONS:
Biological: VAX125 — Single intramuscular dose
  Other Names: STF2.HA1(SI)

SUMMARY:
Is VAX125 safe at doses ranging from 0.1 to 8 ug when delivered i.m. in a single dose regimen Is VAX125 able to induce a post-vaccination serum HAI antibody response in healthy adults against the influenza A virus H1 HA.

DETAILED DESCRIPTION:
Part I: Intramuscular (i.m.) vaccination of a single dose of 0.1 µg, 0.3 µg, 1 µg, 2 µg, 3 µg, 5 µg and 8 µg of STF2.HA1 (SI) (VAX125) to be given on Day 0

Part II: Intramuscular (i.m.) vaccination of a single dose of placebo or one of two dose levels of STF2.HA1 (SI) (VAX125) (optimum dose levels to be determined from the safety and immunogenicity data from Part I of this study) to be given on Day 0

Part I Primary: To assess the safety, reactogenicity, and tolerability of the VAX125 vaccine delivered i.m. in a single dose regimen of dose levels of 0.1 µg, 0.3 µg, 1 µg, 2 µg, 3 µg, 5 µg, and 8 µg in healthy adults 18 - 49 years of age, inclusive.

Secondary: To assess the immunogenicity of the VAX125 vaccine delivered i.m. in a single dose regimen at dose levels of 0.1 µg, 0.3 µg, 1 µg, 2 µg, 3 µg, 5 µg, and 8 µg, for inducing a post-vaccination serum HAI antibody response in healthy adults against the influenza A virus H1 HA.

Part II Primary: To assess the safety, reactogenicity, and tolerability of a single dose of the VAX125 vaccine delivered i.m. in one of two dose levels as compared to placebo, (optimum dose levels to be determined from the safety and immunogenicity data from Part I of this study), in healthy adults 18- 49 years of age, inclusive.

Secondary: To assess the immunogenicity of a single dose the VAX125 vaccine delivered i.m. in one of two dose levels as compared to placebo (optimum dose levels to be determined from the safety and immunogenicity data from Part I of this study) for inducing a post-vaccination serum HAI antibody response in healthy adults against the influenza A virus H1 HA antigen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 49 years inclusive
* Give written informed consent to participate.
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations
* Females should willing to use another reliable form of contraception approved by the Investigator and a negative urine pregnancy test within 24 hours preceding receipt of vaccination
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.

Exclusion Criteria:

* Presence of significant uncontrolled medical or psychiatric illness (acute or chronic). This includes institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed on Day 0 prior to vaccination.
* Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies.
* Cancer, or treatment for cancer, within 3 years. (Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible), excluding basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) which is allowed, unless at vaccination site.
* Impaired immune responsiveness (of any cause), including diabetes mellitus.
* Documented influenza infection with a positive culture in the 6 months prior to screening.
* Presently receiving or history of receiving any medications or treatments that affects the immune system such as allergy shots, immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months prior to screening. Inhaled and topical corticosteroids will be allowed.
* Receipt or planned administration of a nonstudy vaccine within 30 days prior to vaccination and during the study, including licensed influenza vaccines. Immunization on an emergency basis with Tetanus Toxoid Adsorbed for adult use (Td or Tdap) up to 8 days before or at least 8 days after a dose of study vaccine will be allowed. Administration of study vaccine injection can be delayed if a nonstudy vaccine has been administered and will be given as soon as acceptable, as described above, provided the vaccine is not administered within two weeks prior to study enrollment.
* History of anaphylactic type reaction to injected vaccines.
* History of drug or chemical abuse in the year before the study.
* Receipt of any investigational product or nonregistered drug within the 30 days prior to vaccination or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing study period.
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the study period.
* Donation of blood or blood products within 8 weeks prior to vaccination or at any time during the study.
* Acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination; for example, those requiring an absence from work) with or without fever, or a fever >37.9ºC orally. Study vaccine can be administered to persons with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade febrile illness. Vaccination can be delayed until the subject has recovered.
* Any condition that, in the opinion of the investigator, might interfere with study objectives

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, laboratory tests and AEs. | 6 months

SECONDARY OUTCOMES:
Immunogenicity after single intramuscular dose ranging from 0.1 ug to 8 ug for inducing a post-vaccination serum HAI antibody response in healthy adults against the influenza A virus H1 HA antigen. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John J Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Song L, Nakaar V, Kavita U, Price A, Huleatt J, Tang J, Jacobs A, Liu G, Huang Y, Desai P, Maksymiuk G, Takahashi V, Umlauf S, Reiserova L, Bell R, Li H, Zhang Y, McDonald WF, Powell TJ, Tussey L. Efficacious recombinant influenza vaccines produced by high yield bacterial expression: a solution to global pandemic and seasonal needs. PLoS One. 2008 May 21;3(5):e2257. doi: 10.1371/journal.pone.0002257. PMID 18493310
- [Derived] Treanor JJ, Taylor DN, Tussey L, Hay C, Nolan C, Fitzgerald T, Liu G, Kavita U, Song L, Dark I, Shaw A. Safety and immunogenicity of a recombinant hemagglutinin influenza-flagellin fusion vaccine (VAX125) in healthy young adults. Vaccine. 2010 Dec 6;28(52):8268-74. doi: 10.1016/j.vaccine.2010.10.009. Epub 2010 Oct 20. PMID 20969925